CLINICAL TRIAL: NCT01062932
Title: Cycloserine Enhancement of Extinction Learning
Brief Title: Investigation of Cycloserine as a Smoking Cessation Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: H-23305; R21DA023588 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Nicotine Addiction
Keywords: Cycloserine; Nicotine; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cycloserine (Active Comparator)
  Interventions: Drug: Cycloserine

INTERVENTIONS:
Drug: Cycloserine — Oral administration of cycloserine medication (50 mg administered prior to each exposure treatment) on Day 1, 4, 7, and 10 of the study
  Other Names: d-cycloserine; Seromycin
  Arms: Cycloserine
Drug: Placebo — Oral administration of matching placebo pill on Days 1, 4, 7, and 10
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Psychosocial treatments for drug abuse benefit some patients (Rawson et al 2004), but there is an urgent need for new treatment approaches that can improve treatment outcomes. One new approach involves facilitation of extinction of conditioned responses through the use of d-cycloserine, a partial agonist at the NMDA glycine site. This approach has proved useful for the treatment of several anxiety disorders. For example, treatment with d-cycloserine enhanced the efficacy of behavioral treatments for acrophobia (Ressler et al 2004) and social phobia (Hofmann et al 2006) by enhancing extinction of conditioned fear responses. This suggests that d-cycloserine has potential to enhance the efficacy of behavioral treatments for drug dependence by enhancing extinction of conditioned responses to drug cues. In this Phase I Cutting-Edge Basic Research Awards (CEBRA) application we propose a proof-of-concept study to examine effects of treatment with d-cycloserine for facilitating extinction of craving provoked by exposure to cigarette smoking cues. The benefits of this treatment approach together with cognitive behavioral treatment for reducing cigarette smoking will then be determined. Smoking cues will be presented using an established virtual reality simulator(Bordnick et al 2004; Bordnick et al 2005a)

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Want to participate in a treatment aimed at helping them stop smoking cigarettes
* Be English-speaking volunteers between 18-55 years of age
* Meet DSM-IV TR criteria for current nicotine dependence and smoke >10 cigarettes per day for the past year
* Meet DSM-IV TR criteria for cocaine dependence, but not seeking treatment for cocaine dependence at the time of study
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator

Exclusion Criteria:

* Meet DSM-IV TR criteria for abuse or dependence on alcohol or other drugs, except for nicotine and cocaine
* Have psychiatric disorders, such as: current major depression as assessed by SCID; lifetime history of schizophrenia, other psychotic illness, or bipolar illness as assessed by SCID; current organic brain disease or dementia assessed by clinical interview; history of or any current psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; history of seizure disorder or severe head injury
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
* Be pregnant or nursing. Female participants must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry and at the end of study participation
* Have no history of adverse response to d-cycloserine
* Have any other illness, condition, or use of medications, which in the opinion of the P.I. and/or the admitting physician would preclude safe and/or successful completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The effects of four weeks of single dose treatment with d-cycloserine or placebo on craving elicited by exposure to "virtual reality" smoking cues
  The study will evaluate the effects of treatment with d-cycloserine (50mg administered prior to each exposure treatment) or placebo (n=20 per cell), on the efficacy exposure therapy using a virtual reality cue for smoking cessation when combined with cognitive behavioral therapy (CBT). Craving ratings will be assessed using standard questionnaires, which will be completed prior to and following virtual reality cue exposure. Smoking cessation and cocaine use will be assessed at three follow-up visits.

SECONDARY OUTCOMES:
The effects of four weeks of single dose treatment with d-cycloserine or placebo, exposure to virtual reality smoking cues, and provision of manual-driven cognitive behavioral treatment on frequency of cigarette smoking and cocaine use
  Study sessions will include assessment of urinary cocaine and breath CO, and participants will self-report cigarette smoking and cocaine use over the previous week. Smoking cessation and cocaine use will also be assessed at three follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States